CLINICAL TRIAL: NCT07137208
Title: Bilevel Erector Spinae Plane Block Versus Transversus Abdominis Plane Block for Analgesia After Cesarean Delivery Under Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: Bilevel Erector Spinae Plane Block Versus Transversus Abdominis Plane Block for Analgesia After Cesarean Delivery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amany Hazem abdelmaksood EL-deeb, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bilevel ESPB for CS analgesia
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section Wound
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Randomized controlled, single-blind study.
Who Masked: Outcomes Assessor
Masking Description: A single investigator will handle eligibility screening, informed consent, and baseline data collection. An anesthesiology resident, not involved in the study, will administer the spinal anesthesia, record intraoperative data, and prepare the block solution. The patients will be separated from the surgical field and the operators by a large opaque screen. After achieving an upper sensory level of T6 or higher, the primary investigator (who will not participate in anesthesia or postoperative care) will open group allocation envelopes and perform the block after skin closure. All blocks will be done by the same anesthesiologist. Postoperative data will be collected by independent assessors.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilevel ESP block group (Active Comparator): Ultrasound-guided bilevel ESP block will be performed under strict aseptic precautions and patients will be positioned in the right lateral position.
  Interventions: Procedure: ESP block; Drug: Bupivacaine injection
- Posterior TAP block group (Active Comparator): Ultrasound-guided posterior TAP block will be performed under strict aseptic precautions and patients will be positioned the supine position.
  Interventions: Procedure: TAP Block; Drug: Bupivacaine injection

INTERVENTIONS:
Procedure: ESP block — In the ESP group, patients will be positioned in the right lateral position. The ultrasound probe will be placed vertically about 3 cm lateral to the spinous process of T9 to visualize the transverse process, trapezius, and erector spinae muscles. A 22-gauge spinal needle will be inserted in-plane in the cranial-to-caudal direction until the needle tip reaches the fascial plane between the erector spinae muscle and transverse process. Following hydrodissection with 2 mL of sterile saline to confirm needle placement, and negative aspiration to rule out intravascular placement, the local anesthetic will be injected. Likewise, the same block procedure will be performed at the T11 level and on both levels on the other side, 10 mL will be injected at each of the four injection sites.
  Arms: Bilevel ESP block group
Procedure: TAP Block — In the TAP group, patients will be positioned in the supine position. A posterior approach will be employed, with the ultrasound probe placed transversely on the anterolateral abdominal wall, midway between the costal margin and iliac crest, posterior to the midaxillary line. This will allow visualization of the external oblique, internal oblique, and transversus abdominis muscles. The probe will then be moved posteriorly to identify the tapering of the transversus abdominis muscle toward the quadratus lumborum. A 22-gauge spinal needle will be inserted in-plane from anterior to posterior. Following hydrodissection with 2 mL of sterile saline to confirm needle placement, and negative aspiration to rule out intravascular placement, the local anesthetic will be injected into the plane between the internal oblique and transversus abdominis muscles. Likewise, the same block procedure will be performed on the other side.
  Arms: Posterior TAP block group
Drug: Bupivacaine injection — A total of 20 mL of 0.25 bupivacaine will be administered at each side.
  Other Names: 0.25 bupivacaine

SUMMARY:
Optimizing analgesia after cesarian delivery is an essential element of enhancing maternal recovery.A multimodal analgesic approach incorporating truncal blocks can provide effective pain relief with minimal side effects for both mother and infant.The posterior TAP block may provide enhanced effect due to possible retrograde spread to the paravertebral space.The ESP block has emerged as a valuable component of multimodal pain management, providing effective postoperative analgesia for various surgeries, including cesarean delivery. We hypothesized that the bilevel ESP block will offer superior analgesic efficacy compared to the TAP block and may be a valuable addition to multimodal analgesic regimens targeting opioid use reduction.

DETAILED DESCRIPTION:
Optimizing analgesia after cesarian delivery is an essential element of enhancing maternal recovery, as it supports earlier mobilization, thereby reducing the risk of thromboembolic complications. A multimodal analgesic approach incorporating truncal blocks can provide effective pain relief with minimal side effects for both mother and infant. Epidural or intrathecal administration of morphine is the gold standard for post-cesarean analgesia and forms a cornerstone of multimodal pain management strategies.

In recent years, regional anesthesia techniques are increasingly employed to enhance analgesia and minimize systemic opioid use. These include local anesthetic wound infiltration, ilioinguinal/iliohypogastric nerve blocks, and intraperitoneal anesthetic instillation. Fascial plane blocks such as transversus abdominis plane (TAP), quadratus lumborum (QL), and erector spinae plane (ESP) blocks are also employed to target both somatic and visceral pain effectively.The TAP block is widely used for post-cesarean pain relief by blocking the anterior rami of spinal nerves supplying the abdominal wall through local anesthetic spread between the internal oblique and transversus abdominis muscles. While it offers effective somatic analgesia, it lacks visceral pain relief. The posterior TAP block may provide enhanced effect due to possible retrograde spread to the paravertebral space.The ESP block has emerged as a valuable component of multimodal pain management, providing effective postoperative analgesia for various surgeries, including cesarean delivery. It primarily targets the dorsal rami, with potential spread to the ventral rami through paravertebral space, offering broad and segmental analgesic coverage. The block's simplicity, safety, and opioid-sparing effects especially in low thoracic applications have contributed to its growing use in abdominal surgeries.Although early research suggests that the ESP block may reduce pain and opioid consumption following cesarean delivery, conclusive evidence of its superiority over the TAP block is still lacking. Therefore, this study aims to compare the analgesic efficacy of TAP and bilevel ESP blocks in patients undergoing cesarean delivery under spinal anesthesia.

Aim of the study:

This study aims to compare the bilateral bilevel ESP block with the bilateral TAP block for analgesia after cesarean delivery performed under spinal anesthesia.

Sample Size Calculation:

The sample size is determined based on pilot study on 10 patients, which reported a mean ± standard deviation of cumulative fentanyl consumption at 24 hours as 45 ± 28μg. Assuming a two-tailed Student's t-test with a significance level (α) of 0.05 and a power (1-β) of 90%, and targeting an effect size of 0.71, it was calculated that 43 participants per group would be needed to detect a 20-μg reduction in mean cumulative fentanyl consumption-considered the minimal clinically significant difference. To account for potential dropouts, 45 participants will be allocated to each group.

Methods The study will be conducted on healthy parturients with singleton pregnancy scheduled for elective cesarean delivery via a Pfannenstiel incision under spinal anesthesia at the Obstetric Department of Mansoura University Hospitals All the participants will provide written informed consent. The study subjects will be randomly assigned to 2 equal groups (TAP and bilevel ESP groups).

Randomization will be done using the permuted block randomization method. The group allocation codes will be concealed in sequentially numbered, opaque, sealed envelopes which will be opened only after assessing eligibility and obtaining consent.

A single investigator will handle eligibility screening, informed consent, and baseline data collection. An anesthesiology resident, not involved in the study, will administer the spinal anesthesia, record intraoperative data, and prepare the block solution. The patients will be separated from the surgical field and the operators by a large opaque screen. After achieving an upper sensory level of T6 or higher, the primary investigator (who will not participate in anesthesia or postoperative care) will open group allocation envelopes and perform the block after skin closure. All blocks will be done by the same anesthesiologist. Postoperative data will be collected by independent assessors.

Following standard hospital protocol, a pre-anesthetic evaluation will be conducted, Eligible subjects will be instructed to fast from solid food for 8 hours before surgery, while clear fluids will be permitted up to 2 hours before the procedure. An18-gauge IV cannula will be inserted in a large forearm vein.

Study participants will enter the operating room without receiving any premedication. Upon arrival, a standard monitor (electrocardiography, pulse oximetry, and noninvasive blood pressure) will be initiated.

Strict aseptic technique will be used to perform spinal anesthesia in the sitting position at either the L3-L4 or L4-L5 interspace using a 25-gauge spinal needle. Each patient will receive 2.5 mL of 0.5% hyperbaric bupivacaine (12.5 mg) combined with (15 μg) of fentanyl. Surgery will commence once a sensory block at the T6 level or higher is confirmed via pinprick test. If the sensory level remains below T6 after 20 minutes, the spinal anesthesia will be deemed unsuccessful, and the patient will be excluded from the study.

The upper sensory level will be evaluated using a pinprick test 30 minutes after the intrathecal injection and documented accordingly. If the patient experiences abdominal pain or discomfort after surgery begins, 2 mg of IV midazolam will be given. Should the discomfort persist despite midazolam, IV fentanyl and/or propofol will be administered as needed, and the patient will be excluded from the study.

Immediately following the intrathecal injection, the parturients will be placed in a supine position with a 15° left lateral tilt. A 1000 mL bolus of Ringer acetate will be infused over 10 minutes. In all cases, a lower segment cesarean delivery will typically be performed using a Pfannenstiel incision, with exteriorization of the uterus as part of the surgical technique. After fetal delivery, 10 units of oxytocin diluted in 500 mL of Ringer acetate will be administered over 30 minutes.

Throughout the cesarean procedure, continuous monitoring of mean arterial pressure and heart rate will be conducted. If systolic blood pressure drops by 20% from baseline or falls below 90 mmHg, 5 mg of IV ephedrine will be given. If the heart rate decreases to 50 bpm or lower, 0.5 mg of IV atropine will be administered.

The spinal level will be assessed and documented prior to the administration of either type of block.

At the end of surgery, with the patient under full monitoring, either ESP block or TAP block will be performed under ultrasound guidance. A total of 20 mL of 0.25 bupivacaine will be administered at each side.

All women will be instructed to report any symptoms of local anesthetic toxicity, such as circumoral or tongue numbness, visual or auditory disturbance, dizziness, or tinnitus.

Then, women will be transferred to the postoperative anesthesia care unit for routine monitoring and exclusion of acute complications from the blocks, and later to the obstetric department.

In the obstetric department, all the study subjects will receive postoperative standard analgesia, which includes (30 mg of IV ketorolac every 8 hours starting immediately after surgery and 1 gm of IV paracetamol every 8 hours starting 4 hours after surgery).

Rescue analgesia or first postoperative analgesia (fentanyl 25 μg intravenously) will be considered when VAS ≥4 will be observed or upon patient demand with maximum 4-hour dose limit 200 μg.

Statistical analysis:

Statistical analyses will be conducted using SPSS software (version 26). Data normality will be assessed using histograms and the Kolmogorov-Smirnov test. Continuous variables with a normal distribution will be expressed as mean ± standard deviation (SD) and analyzed using the Student's t-test. Non-normally distributed data will be presented as median (range) and compared using the Mann-Whitney U test. Bonferroni correction will be applied to adjust for multiple comparisons. Categorical variables will be presented as number (percentages) and analyzed using the Chi-square test or Fisher's exact test. A two-tailed p-value <0.05 will be considered statistically significant, with a 95% confidence interval. Time to first fentanyl dose will be analyzed using Kaplan-Meier survival analysis and compared using the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Parturients with full term singleton pregnancy.
* American Society of Anesthesiologists (ASA) physical status II.

Exclusion Criteria:

* Body mass index (BMI) ≥ 35 kg/m².
* Cerebrovascular, cardiovascular, hepatic, or renal disease.
* Any contraindication to spinal anesthesia, local anesthetic or opioids.
* Pre-existing chronic pain syndrome or history of recent opioid exposure.
* Inability to comprehend or participate in pain scoring system.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant with singleton full term
Enrollment: 90 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Total analgesic requirements of fentanyl | Up to 24 hours after the procedure
  The amount of fentanyl consumption given as a rescue analgesia to patients will be measured all over the 24 hours.

SECONDARY OUTCOMES:
the first analgesic request time | Up to 24 hours after the procedure
  The time of the first analgesic request for fentanyl will be recorded.
The intensity of postoperative pain | Up to 24 hours after the procedure
  using an 11-point NRS (0 = no pain and 10 = the worst possible pain), both at rest and during movement (e.g., lower limb flexion and extension, trunk movement by turning from a supine position to either the right or left side, and coughing) at 2, 4, 6, 12, and 24 hours postoperatively, considering the time of completion of the respective block procedure (i.e., deposition of the required amount of local anesthetic into the desired plane) on each side as "time 0."
Patient satisfaction | Up to 24 hours after the procedure
  Patient satisfaction with postoperative analgesia will be assessed at 24 hours using a 5-point scale (1 = very unsatisfied, 2 = unsatisfied, 3 = fair, 4 = satisfied, and 5 = very satisfied).
Incidence of any adverse effects | Up to 24 hours after the procedure
  Any adverse effects (nausea, vomiting, drowsiness, itching, pruritus) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Amany H Eldeeb, Principal Investigator — Faculty of Medicine, Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamel AAF, Amin OAI, Ibrahem MAM. Bilateral Ultrasound-Guided Erector Spinae Plane Block Versus Transversus Abdominis Plane Block on Postoperative Analgesia after Total Abdominal Hysterectomy. Pain Physician. 2020 Jul;23(4):375-382. PMID 32709172
- [Result] Eksteen A, Wagner J, Kleyenstuber T, Kamerman P. Comparison of erector spinae plane and transversus abdominis plane block for postoperative analgesia after caesarean delivery under spinal anaesthesia: A randomised controlled trial. Int J Obstet Anesth. 2024 Nov;60:104259. doi: 10.1016/j.ijoa.2024.104259. Epub 2024 Aug 30. PMID 39307664
- [Result] Chin KJ, El-Boghdadly K. Mechanisms of action of the erector spinae plane (ESP) block: a narrative review. Can J Anaesth. 2021 Mar;68(3):387-408. doi: 10.1007/s12630-020-01875-2. Epub 2021 Jan 6. PMID 33403545
- [Result] Canakci E, Gultekin A, Cebeci Z, Hanedan B, Kilinc A. The Analgesic Efficacy of Transverse Abdominis Plane Block versus Epidural Block after Caesarean Delivery: Which One Is Effective? TAP Block? Epidural Block? Pain Res Manag. 2018 Oct 17;2018:3562701. doi: 10.1155/2018/3562701. eCollection 2018. PMID 30416635
- [Result] Silverman M, Zwolinski N, Wang E, Lockwood N, Ancuta M, Jin E, Li J. Regional Analgesia for Cesarean Delivery: A Narrative Review Toward Enhancing Outcomes in Parturients. J Pain Res. 2023 Nov 10;16:3807-3835. doi: 10.2147/JPR.S428332. eCollection 2023. PMID 38026463
- [Result] Hussain N, Brull R, Thaete L, Fuller S, D'Souza RS, Mankinen-Abdallah Y, Essandoh MK, Weaver TE, Abdallah FW. The analgesic effects of novel fascial plane blocks compared with intrathecal morphine after Caesarean delivery: a systematic review and meta-analysis. Br J Anaesth. 2025 May;134(5):1415-1431. doi: 10.1016/j.bja.2025.01.032. Epub 2025 Mar 11. PMID 40074621
- [Result] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Result] Mitchell KD, Smith CT, Mechling C, Wessel CB, Orebaugh S, Lim G. A review of peripheral nerve blocks for cesarean delivery analgesia. Reg Anesth Pain Med. 2019 Oct 25:rapm-2019-100752. doi: 10.1136/rapm-2019-100752. Online ahead of print. PMID 31653797
- [Result] Sangkum L, Tangjitbampenbun A, Chalacheewa T, Brennan K, Liu H. Peripheral Nerve Blocks for Cesarean Delivery Analgesia: A Narrative Review. Medicina (Kaunas). 2023 Nov 4;59(11):1951. doi: 10.3390/medicina59111951. PMID 38004000